CLINICAL TRIAL: NCT04581018
Title: An Evaluation of a Synbiotic Formula for Symptom Improvement in Hospitalised Patients With COVID-19 Infection
Brief Title: An Evaluation of a Synbiotic Formula for Patients With COVID-19 Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Siew Chien NG (Other)
Responsible Party: Sponsor-Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Synbiotic COV study
Record Dates: First submitted 2020-08-11; First posted 2020-10-09 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Covid19; Microbiota
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health supplements + standard care (Active Comparator): 28 days of health supplements (Synbiotic) daily plus standard care
  Interventions: Other: Health supplements
- Standard care (No Intervention): No intervention

INTERVENTIONS:
Other: Health supplements — 28 days of health supplements (synbiotic), 4g daily
  Arms: Health supplements + standard care

SUMMARY:
In December 2019, a cluster of pneumonia cases of unidentified cause emerged in Wuhan,was identified as the culprit of this disease currently being identified as "Coronavirus Disease 2019" (COVID-19) by World Health Organization.

Coronavirus was found to not only target the patient's lungs but also multiple organs. Around 2-33% of Coronavirus Disease-19 patients developed gastrointestinal symptoms. Studies have shown that Severe acute respiratory syndrome coronavirus 2 (SAR-CoV-2) was found in patient's feces, suggesting that the virus can spread through feces. In our previous study, stool samples from 15 patients with COVID-19 were analysed. Depleted symbionts and gut dysbiosis were noted even after patients were detected negative of SARS-CoV-2. A series of microbiota were correlated inversely with the disease severity and virus load. Gut microbiota could play a role in modulating host immune response and potentially influence disease severity and outcomes.

The investigators are uncertain about the impact of synbiotic on patients with COVID-19. However, a therapeutic strategy aiming at investigating the gut Imicrobiota of patients with COVID-9 who take synbiotic or not, leading to lesser progression to severe disease, less hospital stay and improved quality of life.

DETAILED DESCRIPTION:
In December 2019, a cluster of pneumonia cases of unidentified cause emerged in Wuhan, Hubei province, China. In early January, a novel betacoronavirus forming another clade within the subgenus sarbecovirus, now named SARS-CoV-2, was identified as the culprit of this disease currently being identified as "Coronavirus Disease 2019" (COVID-19) by WHO.

Coronavirus was found to not only target the patient's lungs, but also multiple organs. Around 2-33% of COVID-19 patients developed gastrointestinal symptoms. Studies have shown that SAR-CoV-2 was found in patient's feces, suggesting that the virus can spread through feces. In our previous study, stool samples from 15 patients with COVID-19 were analysed. Depleted symbionts and gut dysbiosis were noted even after patients were detected negative of SARS-CoV-2. A series of microbiota were correlated inversely with the disease severity and virus load. Gut microbiota could play a role in modulating host immune response and potentially influence disease severity and outcomes.

In July 2020, there are more than 15 million confirmed cases globally with 620 thousand deaths. Currently, there are more than 2000 confirmed cases of COVID-19 in Hong Kong. The investigators are uncertain about the impact of synbiotic on patients with COVID-19. However, a therapeutic strategy aiming at investigating the gut Imicrobiota of patients with COVID-9 who take synbiotic or not, leading to lesser progression to severe disease, less hospital stay and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or above; and
2. A confirmed diagnosis of SARS-CoV-2 infection using the PCR according to the standard of according to Centre for Health Protection, Department of Health, HK at recruitment and that require admission to the hospitalization area; and
3. Written informed consent is obtained

Exclusion Criteria:

1. Subjects admitted to Intensive Care Unit or on ventilator
2. Known allergy or intolerance to the intervention product or its components
3. Any known medical condition that would prevent taking oral probiotics or increase risks associated with probiotics including but not limited to inability to swallow/aspiration risk and no other methods of delivery (e.g no G/J tube)
4. Known increased infection risk due to immunosuppression such as:

   * Prior organ or hematopoietic stem cell transplant
   * Neutropenia (ANC <500 cells/ul)
   * HIV and CD4 <200 cells/ul
5. Known history or active endocarditis
6. Recent on CAPD or hemodialysis-
7. Documented pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Combined symptom score | 4 weeks
  Combined symptom score improvement of the first 4 weeks. Symptoms score assessment ranges from 20-80. The higher the score, the worse the symptoms.

SECONDARY OUTCOMES:
Clinical improvement | 4 weeks
  Compare the number and severity of symptoms existing by checking the list in symptoms assessment such as cough, shortness of breath, fever and gastrointestinal symptoms like anorexia, nausea, vomiting, abdominal pain, bloating before and during the study
Time to develop antibody against SARS-CoV-2 | 16 days
  Compare the time to develop antibody against SARS-CoV-2 in both group
Quality of life measured by EQ-5D-5L | 4 weeks
  Improvement of quality of life measured by EQ-5D-5L. EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.The index can be calculated by deducting the appropriate weights from 1, the value for full health (i.e. state 11111). Each category ranges from 1 to 5. The small the number, the better the health. The EQ-VAS is a vertical visual analogue scale that ranges 0-100 (higher score indicates better imaginable health).
Quality of life measured by SF-12 | 4 weeks
  Improvement of quality of life measured by SF-12. SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. There are formulas for transformation of scale scores so that they will range from 0-100. High score in functioning items indicates better functioning while high score in pain items indicates freedom from pain.
Duration of hospital stay | up to 3 months
  Measure the duration of hospital stay in both group
Time to negative PCR | through study completion, an average of 1 year
  Compare the time to negative PCR in both group
Trend of symptom score | 4 weeks
  Trend of symptom score, ranges from 26-104. The higher the score, the worse the symptoms.
Gastrointestinal symptoms | 4 weeks
  Duration of gastrointestinal symptoms such as anorexia, nausea, vomiting, abdominal pain, bloating within 4 week.
Changes in fecal bacteria metabolites | weeks 2, 4, 5 and 8 months 3, 6, 9 and 12
  Changes in fecal bacteria metabolites measured by PCR at different time points
Change in plasma cytokines level | week 2 and week 5
  Change in plasma cytokines level at week 2 and week 5 compared with baseline
Changes in the gut microbiome | weeks 1, 2, 3, 4, 5, 8 and months 3, 6, 9 and 12
  Changes in the gut microbiome (bacteria, virome and fungome) measured by metagenomics at different time points (weeks 1, 2, 3, 4, 5 and months 3, 6, 9 and 12) compared to baseline
Number of admission to Intensive Care Unit | 4 weeks
  Number of admission to Intensive Care Unit
Number of subjects with home discharge | 4 weeks
  Number of subjects with home discharge
Number of mortality | 4 weeks
  Number of mortality
Number of days absent from work | 3 months
  Number of days absent from work since admission
Change of quality of life questionnaire | week 8, months 3, 6, 9 and 12
  Change in score on Quality of life using EQ-5D-5L and SF-12. EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.The index can be calculated by deducting the appropriate weights from 1, the value for full health (i.e. state 11111). Each category ranges from 1 to 5. The small the number, the better the health. The EQ-VAS is a vertical visual analogue scale that ranges 0-100 (higher score indicates better imaginable health). While the SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. There are formulas for transformation of scale scores so that they will range from 0-100. High score in functioning items indicates better functioning while high score in pain items indicates freedom from pain.
Number of adverse event | 3 months
  Number of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Wong CK, Lam CW, Wu AK, Ip WK, Lee NL, Chan IH, Lit LC, Hui DS, Chan MH, Chung SS, Sung JJ. Plasma inflammatory cytokines and chemokines in severe acute respiratory syndrome. Clin Exp Immunol. 2004 Apr;136(1):95-103. doi: 10.1111/j.1365-2249.2004.02415.x. PMID 15030519
- [Background] Holshue ML, DeBolt C, Lindquist S, Lofy KH, Wiesman J, Bruce H, Spitters C, Ericson K, Wilkerson S, Tural A, Diaz G, Cohn A, Fox L, Patel A, Gerber SI, Kim L, Tong S, Lu X, Lindstrom S, Pallansch MA, Weldon WC, Biggs HM, Uyeki TM, Pillai SK; Washington State 2019-nCoV Case Investigation Team. First Case of 2019 Novel Coronavirus in the United States. N Engl J Med. 2020 Mar 5;382(10):929-936. doi: 10.1056/NEJMoa2001191. Epub 2020 Jan 31. PMID 32004427
- [Background] Yeo C, Kaushal S, Yeo D. Enteric involvement of coronaviruses: is faecal-oral transmission of SARS-CoV-2 possible? Lancet Gastroenterol Hepatol. 2020 Apr;5(4):335-337. doi: 10.1016/S2468-1253(20)30048-0. Epub 2020 Feb 20. No abstract available. PMID 32087098
- [Background] Liang W, Feng Z, Rao S, Xiao C, Xue X, Lin Z, Zhang Q, Qi W. Diarrhoea may be underestimated: a missing link in 2019 novel coronavirus. Gut. 2020 Jun;69(6):1141-1143. doi: 10.1136/gutjnl-2020-320832. Epub 2020 Feb 26. No abstract available. PMID 32102928
- [Background] Hashimoto T, Perlot T, Rehman A, Trichereau J, Ishiguro H, Paolino M, Sigl V, Hanada T, Hanada R, Lipinski S, Wild B, Camargo SM, Singer D, Richter A, Kuba K, Fukamizu A, Schreiber S, Clevers H, Verrey F, Rosenstiel P, Penninger JM. ACE2 links amino acid malnutrition to microbial ecology and intestinal inflammation. Nature. 2012 Jul 25;487(7408):477-81. doi: 10.1038/nature11228. PMID 22837003
- [Background] Zuo T, Zhan H, Zhang F, Liu Q, Tso EYK, Lui GCY, Chen N, Li A, Lu W, Chan FKL, Chan PKS, Ng SC. Alterations in Fecal Fungal Microbiome of Patients With COVID-19 During Time of Hospitalization until Discharge. Gastroenterology. 2020 Oct;159(4):1302-1310.e5. doi: 10.1053/j.gastro.2020.06.048. Epub 2020 Jun 26. PMID 32598884
- [Background] WHO Coronavirus Disease (COVID-19) Dashboard. [Assessed on 24 Jul 2020]. https://covid19.who.int/
- [Background] Latest situation of cases of COVID-19. [Assessed on 24 Jul 2020]. https://www.chp.gov.hk/files/pdf/local_situation_covid19_en.pdf
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Docherty AB, Harrison EM, Green CA, Hardwick HE, Pius R, Norman L, Holden KA, Read JM, Dondelinger F, Carson G, Merson L, Lee J, Plotkin D, Sigfrid L, Halpin S, Jackson C, Gamble C, Horby PW, Nguyen-Van-Tam JS, Ho A, Russell CD, Dunning J, Openshaw PJ, Baillie JK, Semple MG; ISARIC4C investigators. Features of 20 133 UK patients in hospital with covid-19 using the ISARIC WHO Clinical Characterisation Protocol: prospective observational cohort study. BMJ. 2020 May 22;369:m1985. doi: 10.1136/bmj.m1985. PMID 32444460
- [Background] Janowitz T, Gablenz E, Pattinson D, Wang TC, Conigliaro J, Tracey K, Tuveson D. Famotidine use and quantitative symptom tracking for COVID-19 in non-hospitalised patients: a case series. Gut. 2020 Sep;69(9):1592-1597. doi: 10.1136/gutjnl-2020-321852. Epub 2020 Jun 4. PMID 32499303
- [Derived] Liang JQ, Zeng Y, Lau EYT, Sun Y, Huang Y, Zhou T, Xu Z, Yu J, Ng SC, Chan FKL. A Probiotic Formula for Modulation of Colorectal Cancer Risk via Reducing CRC-Associated Bacteria. Cells. 2023 Apr 25;12(9):1244. doi: 10.3390/cells12091244. PMID 37174650